CLINICAL TRIAL: NCT01027481
Title: Response of Retinal Vessels to Anti Vascular Endothelial Growth Factor (VEGF) Treatment in Patients With Branch Retinal Vein Occlusion (BRVO)
Brief Title: Ranibizumab in Patients With Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Stefan Sacu, Ass. Professor, Department of Ophthalmology, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2007-11

CONDITIONS: Retinal Vein Occlusion
Keywords: lucentis, macular edema, branch retinal vein occlusion
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lucentis — intravitreally administration of 0.05 ml Lucentis
  Other Names: RANIBIZUMAB (Lucentis 0.05 ml, Novartis)

SUMMARY:
In a recent study we could show that the early retinal venous vasoconstriction after grid photocoagulation in branch retinal vein occlusion (BRVO) is closely correlated to the visual outcome after three months. This could be of clinical importance, because the degree of vasoconstriction might be an early marker of treatment success, compatible with the idea that hypoxia is the major trigger of VEGF in BRVO. The present study evaluates the response of retinal vessel diameters to anti VEGF treatment with lucentis in patients with BRVO. This is done in an effort to gain insight into the retinal hemodynamic consequences of anti VEGF treatment in BRVO. The hypothesis that anti VEGF treatment is associated with a vasoconstrictor response in retinal vessel in patients with BRVO is tested.

DETAILED DESCRIPTION:
To investigate the response of retinal vessel diameters to lucentis treatment in patients with BRVO and to correlate these changes with changes in functional outcome after 3 months.

Pilot study in patients scheduled for intravitreal anti-VEGF (Lucentis™) treatment with BRVO

30 patients with BRVO scheduled for intravitreal anti-VEGF treatment Intravitreous administration of Ranibizumab (Lucentis ™)

Main outcome measure: Retinal vessel diameters

Secondary outcome measures: Retrobulbar flow velocities, best-corrected visual acuity, macular sensitivity assessed with Microperimetry, objective functional response assessed with mfERG, anatomic changes in the macula region as assessed with StratusOCT and prototype of a Cirrus-OCT(which is available at the Department of Ophthalmology, Medical University of Vienna), angiographical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* male or female, at least 18 years of age.
* ophthalmoscopic evidence of recent BRVO, that is, a history of 3 months.
* macular edema secondary to BRVO in the study eye scheduled for intravittreal anti-VEGF as primary treatment.
* retinal thickness of > 300 µm by OCT in the central subfield of the study eye at baseline.
* VA decrease attributable to the edema.
* written informed consent has been obtained.
* female patients of childbearing potential must have a negative urine pregnancy test.

Exclusion Criteria:

* Uncontrolled sytemic disease
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Any ocular condition that in the opinion of the investigator would prevent a 15-letter improvement in visual acuity (eg severe macular ischemia)
* History of glaucoma, aphakie or presence of anterior chamber intraocular lens, active reinal neovascularisation, choroidal neovascularisation, significant cataract, presence of rubeosis iridis, any ocular infection, history of pars plana vitrectomy, anticipated need for ocular surgery in the study eye during the study perios.
* contraindication to pupil dilation known allergy or contraindication to the use of fluorescein.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Main outcome measure: Retinal vessel diameters | weeks 1, 4 and 16

SECONDARY OUTCOMES:
Secondary outcome measures: Retrobulbar flow velocities, best-corrected visual acuity, macular sensitivity, objective functional response, anatomic changes in the macula region, angiographical outcomes. | weeks 1,4 and16

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sacu, Ass. Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Vienna General Hospital, Vienna, Austria

REFERENCES:
- [Derived] Sacu S, Pemp B, Weigert G, Matt G, Garhofer G, Pruente C, Schmetterer L, Schmidt-Erfurth U. Response of retinal vessels and retrobulbar hemodynamics to intravitreal anti-VEGF treatment in eyes with branch retinal vein occlusion. Invest Ophthalmol Vis Sci. 2011 May 9;52(6):3046-50. doi: 10.1167/iovs.10-5842. PMID 21051706